CLINICAL TRIAL: NCT05427032
Title: Improved Health-related Quality of Life During Peptide Receptor Radionuclide Therapy in Patients With Neuroendocrine Tumours
Brief Title: HRQoL During PRRT in Patients With NETs
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: HRQoL PRRT
Record Dates: First submitted 2022-05-13; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Neuroendocrine Tumors; Quality of Life; Peptide Receptor Radionuclide Therapy
Keywords: NETs; PRRT; HRQoL
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuroendocrine tumours (NETs) can arise in different locations in the body, and may give rise to hormonal symptoms, which may affect the patients' health-related quality of life (HRQoL). Up to four cycles of peptide receptor radionuclide therapy (PRRT) have been shown effective for symptom alleviation and prolonging survival. The aim of this study is to assess the patient's perspective, regarding changes in their HRQoL during, and at long-term follow-up after, PRRT. Patients with NET will rate their HRQoL before PRRT cycles one and four, and 1-8 years after PRRT. The patients' HRQoL will be compared to a matched reference population. The investigators hope that this study will reveal specific care needs for patients wiht NET and may provide information that will make it possible to deliver a more person-centered care.

DETAILED DESCRIPTION:
The inclusion criteria for PRRT were tumour somatostatin receptor expression higher than that in the normal liver found on somatostatin receptor scintigraphy (Krenning score 3 and 4), or on 68Ga-DOTATOC positron emission tomography (PET), and sufficient bone marrow, liver and kidney function. DOTATATE was labelled in house with 177Lu (IDB Holland BV, Noord Brabant, Netherlands). Up to nine cycles were given, yet a majority of patients received four cycles of PRRT.

The patients' medical records were reviewed regarding functional status (functioning versus non-functioning tumours), gender, age at diagnosis and at 1st PRRT, marital and employment status, PRRT cycles received, previous treatments and body mass index (BMI).

HRQoL was assessed using the questionnaires for cancer in general, EORTC QLQ-C30, and the gastrointestinal NET-specifically EORTC QLQ-GINET21 at every cycle.

From a large random sample (n=4,910) of the Swedish adult population, a reference population was extracted. They all had chronical diseases (diabetes, cardiac, respiratory, renal or other specified conditions) and were age and gender matched. The reference population completed only the QLQ-C30 questionnaire.

In order to investigate how HRQoL developed during the eight years after PRRT, the questionnaires were sent to 58 patients.

ELIGIBILITY:
Inclusion Criteria:

* Receiving PRRT
* NET diagnosis

Exclusion Criteria:

* Not able to speak and read in Swedish or English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving PRRT at Uppsala University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2009-01-10 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in health related quality of life at cycle 4 | Baseline and before cycle 4 (each cycle is between 28-42 days)
  EORTC QLQ-C30 and QLQ-GINET21 is validated, self-reported instrument assessing health related quality of life during the past week. The instruments are composed of both multi-item scales and singe-items measures. These include five functional scales, three symptom scales, a global health status scale, and six single items.